CLINICAL TRIAL: NCT04701814
Title: The Effect of Biomechanical Scapular Mobilization With Movement and Motor Learning in Shoulder Impingement Patients
Brief Title: The Effect of Biomechanical Scapular Mobilization With Movement and Motor Learning
Acronym: BSMWM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pharos University in Alexandria (Other)
Responsible Party: Principal Investigator, Moataz Abdelaal, Demonstrator in Faculty of Physical Therapy, Pharos University, Alexandria, Egypt., Pharos University in Alexandria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUA 201901013
Record Dates: First submitted 2021-01-05; First posted 2021-01-08 (Actual); Results first posted 2021-04-14 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-04

CONDITIONS: Shoulder Impingement Syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Movement

STUDY DESIGN:
Intervention Model Description: Patients were divided randomly in two equal groups (A and B): Group A (controlled group):
  They were received traditional physical therapy program including: passive range of motion (PROM)/ active assisted range of motion (AAROM)/ active range of motion (AROM), strengthen of rotator cuff, biceps, shoulder and scapular muscles, ultrasound (5 min. - 1.5 W/c.m2 - 1 MHZ), electrical stimulation ( interferential bipolar technique for 20 min. on shoulder joint). Group B (study group): they have received the same physical therapy program as in group A, in addition to Biomechanical scapular mobilization with movement and motor learning.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (controlled group) (Active Comparator): received passive range of motion (PROM)/ active assisted range of motion (AAROM)/ active range of motion (AROM) exercises, strengthen of rotator cuff, biceps, shoulder and scapular muscles, ultrasound (5 min. - 1.5 W/c.m2 - 1 MHZ), electrical stimulation ( interferential bipolar technique for 20 min. on shoulder joint). This treatment was repeated three times per weeks with 24 hours rest for 3 weeks.
  Interventions: Other: biomechanical scapular mobilization with movement and motor learning
- group B(Study group) (Active Comparator): All patients in group B received biomechanical scapular mobilization with movement and motor learning and traditional methods.
  Interventions: Other: biomechanical scapular mobilization with movement and motor learning

INTERVENTIONS:
Other: biomechanical scapular mobilization with movement and motor learning — the therapist applied posterior tilt and exteral rotation with upward rotation mobilization to scapula and therapist also warp bilt around GH joint to applied inferior and posterior glid then ask patient to elevate his arm. then we applied motor learning approach by asking patient to elevate his arm with maintaining of external rotation with posterior glid of scapula.

SUMMARY:
the study about new mobilization technique used in shoulder impingement syndrome patient to increase the range of motion of elevation, decrease the pain, and increasing the function level, this technique is based on normal mechanics that occur inside the joint during certain movement.

DETAILED DESCRIPTION:
The study is about a new technique of mobilization based on normal biomechanics that occurs during the movements of a joint. For example, shoulder abduction or elevation needs the scapula to move upward rotation with posterior tilt and external rotation. Moreover, needs glenohumeral (GH) joint glide inferior and posterior these movements occur normally to permit us to elevate our shoulder without any restriction and the full range of motion(ROM). so in the patients with shoulder problems and have difficulties reaching full ROM of elevation the investigators applied mobilization of scapula toward upward rotation with external rotation and posterior tilt and by using mobilization belt applied posterior and inferior glide to GH joint. However, mobilization techniques have a short-term effect to enhance this effect, the investigators adding a motor learning approach to achieve a long-term effect and prevent recurrent .the investigators applied this technique 3 times per week for 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

clinical diagnosis: shoulder impingement syndrome.

1. History of shoulder pain when they elevated their arm.
2. Limited range of motion due to the pain.
3. Pain localized at the painful point at proximal anterolateral shoulder region or medical diagnosis of shoulder impingement syndrome with at least 2 positive impingement tests including Neer, Hawkins, or Jobe test.

Exclusion Criteria:

* Fibromyalgia.
* Fracture, dislocation, or subluxation of the shoulder.
* history of trauma.
* shoulder surgery.
* numbness or tingling in the upper limb.
* Corticosteroids injection within 1 year.
* systemic illness.
* ligamentous laxity

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2021-10-22 (Actual); Study Completion 2021-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Moataz A. Mohamed, (B.Sc.P.T.), Study Chair — Pharos University in Alexandria
Locations (1):
- Pharos university in Alexandria, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Surenkok O, Aytar A, Baltaci G. Acute effects of scapular mobilization in shoulder dysfunction: a double-blind randomized placebo-controlled trial. J Sport Rehabil. 2009 Nov;18(4):493-501. doi: 10.1123/jsr.18.4.493. PMID 20108851
- Available data/document: Book — http://www.elsevier.com. — Neumann, D. D. (2010). kinesology of musculoskeletal system. In Mosby, Inc., an affiliate of Elsevier Inc. The book described normal biomechanics of the shoulder during the elevation.
- Available data/document: Book — https://doi.org/10.1017/CBO9781107415324.004 — the posterior glid and inferior glid of GH joint is increasing the range of motion and decreasing the pain

RESULTS

PARTICIPANT FLOW:
Groups:
- Group B(Study Group): All patients in group B received same treatment as group A with adding biomechanical scapular mobilization with movement and motor learning.
  biomechanical scapular mobilization with movement and motor learning: the therapist applied posterior tilt and exteral rotation with upward rotation mobilization to scapula and therapist also warp bilt around GH joint to applied inferior and posterior glid then ask patient to elevate his arm. then we applied motor learning approach by asking patient to elevate his arm with maintaining of external rotation with posterior glid of scapula.
Period: Overall Study
Arm/Group | Group A (Controlled Group) | Group B(Study Group)
Started | 20 | 18
Completed | 15 | 15
Not Completed | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Group B(Study Group): All patients in group B received same treatment as group A with biomechanical scapular mobilization with movement and motor learning.
  biomechanical scapular mobilization with movement and motor learning: the therapist applied posterior tilt and exteral rotation with upward rotation mobilization to scapula and therapist also warp bilt around GH joint to applied inferior and posterior glid then ask patient to elevate his arm. then we applied motor learning approach by asking patient to elevate his arm with maintaining of external rotation with posterior glid of scapula.
- Total: Total of all reporting groups
Arm/Group | Group A (Controlled Group) | Group B(Study Group) | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 35.1 (8.123) | 35.3 (7.943) | 35.2 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 5 | 5 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Egypt | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale
Description: 1. Visual Analogue Scale: was used to evaluate the intensity of pain, which The pain VAS is a continuous scale comprised of a horizontal (HVAS) or vertical (VVAS) line, usually, 10 centimetres in length, anchored by 2 verbal descriptors, one for each symptom extreme. For pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 10 centimetres).
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Group B(Study Group): All patients in group B received same treatment as group A but adding biomechanical scapular mobilization with movement and motor learning to treatment.
  biomechanical scapular mobilization with movement and motor learning: the therapist applied posterior tilt and exteral rotation with upward rotation mobilization to scapula and therapist also warp bilt around GH joint to applied inferior and posterior glid then ask patient to elevate his arm. then we applied motor learning approach by asking patient to elevate his arm with maintaining of external rotation with posterior glid of scapula.
Arm/Group | Group A (Controlled Group) | Group B(Study Group)
Number analyzed (Participants) | 15 | 15
score on a scale | 4.2 (1.474) | 0.9 (1.280)

2. Primary Outcome: Universal Goniometer
Description: Universal goniometer: was used to measure the available range of motion at a joint. where used to measure an available range of motion of abduction and flexion of the shoulder joint.
Time Frame: 3 weeks
Measure: Mean (Standard Deviation); unit: Degree
Arm/Group | Group A (Controlled Group) | Group B(Study Group)
Number analyzed (Participants) | 15 | 15
Degree
  Abduction | 85.7 (9.083) | 130.9 (8.302)
  Flexion | 131.7 (10.761) | 173.4 (6.544)

ADVERSE EVENTS:
Time Frame: 5 months
Description: The study isn't including serious adverse events: Adverse events that are not Serious Adverse Events.
  the study is depend on manual therapy that its evidence base to occur any adverse effect is very low may be occur with manipulation technique more than mobilization. when we check the patients after technique to record any adverse events, we found nothing so there is no any adverse event. Also, we have not found any study recorded adverse event due to using mobilization technique in shoulder.
Arm/Group | Group A (Controlled Group) | Group B(Study Group)
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 1/2 | 0/1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (Controlled Group) (N=2) | Group B(Study Group) (N=1)
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — shoulder pain for a day or hours due to overdose of mobilization

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-10-13): https://cdn.clinicaltrials.gov/large-docs/14/NCT04701814/Prot_SAP_ICF_000.pdf